CLINICAL TRIAL: NCT00763399
Title: Phase 4 Study of Probiotics on Intestinal Bacterial Population and Immune Modulation
Brief Title: Effect of Probiotics on Intestinal Bacterial Population and Immune Modulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chang Chen, MD, Department of pediatrics, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 97-0549B
Record Dates: First submitted 2008-09-23; First posted 2008-10-01 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Diarrhea; Constipation
Keywords: probiotics
MeSH Terms: conditions — Diarrhea; Constipation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 97-0549B (Experimental)
  Interventions: Dietary Supplement: probiotics (antibiophilus(Lactobacillus casei), bio-three)

INTERVENTIONS:
Dietary Supplement: probiotics (antibiophilus(Lactobacillus casei), bio-three) — probiotics (antibiophilus(Lactobacillus casei), bio-three) 4x 10^8CFU/day

SUMMARY:
The balance between immunogenic and tolerogenic activities in human immune system strongly depends on microflora-induced pro-and anti-inflammatory activities. Probiotics are important components of microflora. The interactions of the different strains of probiotics and the cells of immune system are largely unknown.

There are many mechanisms by which probiotics enhance intestinal health, including stimulation of immunity, competition for limited nutrients, inhibition of epithelial and mucosal adherence, inhibition of epithelial invasion and production of antimicrobial substances.

Fecal immunoglobulin A(IgA), lactoferrin and calprotectin were determined by enzyme-linked immunosorbent assay(ELISA) and compared in different groups. Other clinical symptoms or signs, including fever, vomiting, diarrhea, abdominal pain, bloating abdomen, daily intake and body weight were also assessed.

The first aim of our study is to evaluate the role of probiotics and their preparation products on the restoration of intestinal bacterial population. The second aim of our study is determining the immunomodulating effects or anti-inflammatory effects of probiotics on the host (human being). We try to seek to gain an advanced understanding of probiotics versus intestinal microorganism and host interactions, as well as mucosal immune responses to probiotics in the intestine.

DETAILED DESCRIPTION:
Some clinical parameters were evaluated according to the following: primary outcome (severity of diarrhea), and secondary outcome including body weight change, appetite and daily intake, bloating or abdominal distension, abdominal pain or colic, constipation, fever, and vomiting were also assessed.

Peripheral blood isolated by Lymphoprep, washed twice in normal saline and once in medium, and suspended in medium [RPMI 1640] to a density of 1 x 106/mL. PBMCs will be isolated from blood donor buffy coats by density gradient centrifugation. The concentration of PBMCs will be adjusted to 106 cells per ml in complete medium, and the cells will be transferred to 24-well plates.Cell surface phenotype expression and intracellular staining. Cells will be stained using a panel of monoclonal antibody (MAb) directed against surface antigens expressed by lymphocytes, monocytes and the appropriate species-specific immunoglobulin G isotype controls. Cells will be acquired using an FACScan (Becton Dickinson) and analyzed with Cell Quest software.

To assess the colonization of intestinal bacteria, fecal samples were collected from each patient on day 0 (the day when patients were enrolled), day 3 and day 7 after probiotics or placebo treatment. The fecal specimens were weighed, homogenized, and serially diluted and plated on selective agar for analysis of bacteria. Fecal bacteria count was expressed as log10 CFU/g feces.

Fecal samples were collected during the treatment period. IgA levels were performed on homogenized fecal samples. Total IgA was determined using goat anti-human IgA-HRP conjugate. The reaction was developed with tetramethyl benzidine (TMB; Zymed Labs.) and read at 450 nm. OD values were converted to ng/g feces of total IgA by comparison with a standard curve developed with anti-human IgA.

The stool samples were prepared and analyzed for lactoferrin. A polyclonal antibody specific for lactoferrin has been pre-coated onto a microplate. Lactoferrin in standards and samples is sandwiched by the immobilized antibody and a biotinylated polyclonal antibody specific for lactoferrin, which is recognized by a streptavidin-peroxidase conjugate. Absorbance is read at OD 450 nm. Lactoferrin was expressed as μg/g feces.

The stool samples were prepared and analyzed for calprotectin. The supernatant was collected and frozen at -20°C. The supernatants were thawed and calprotectin was analyzed with the quantitative calprotectin ELISA and read at OD 450 nm. Calprotectin was expressed as μg/g feces.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea
* constipation

Exclusion Criteria:

* Shock
* Sepsis
* Past history with GI tract surgery
* Immunodeficiency

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea, number of stool passage, bacterial culture for intestinal or cytokine | within 4 weeks

SECONDARY OUTCOMES:
body weight change, appetite and daily intake, Fecal IgA, lactoferrin and calprotectin levels | Within first two weeks
  secondary outcome including body weight change, appetite and daily intake, bloating or abdominal distension, abdominal pain or colic, constipation, fever, and vomiting were also assessed. IgA levels and bacterial culture were performed on homogenized fecal samples. Fecal lactoferrin and calprotectin levels were measured with samples of feces.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Chen, MD, Principal Investigator — Pediatric Department, Chang Gung Memorial Hospital, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan